CLINICAL TRIAL: NCT01463280
Title: Tumescent Lidocaine Effects on Platelet Function Following Liposuction Surgical Trauma: a Prospective Controlled Dosage-response Phase I Clinical Trial
Brief Title: Effect of Tumescent Lidocaine on Platelet Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Klein, Jeffrey A., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Klein-LidoLipo; WIRB Pr#20102004 (Other: Western IRB)
Record Dates: First submitted 2011-09-26; First posted 2011-11-01 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Thromboembolism
Keywords: Platelets; Inhibition; Lidocaine; Thromboembolism; Prevention; Lidocaine effects on platelets
MeSH Terms: conditions — Inhibition, Psychological; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tumescent lidocaine infiltration (Experimental): Assess Platelet function with respect to dosage of tumescent lidocaine There is only one arm.
  Interventions: Drug: tumescent lidocaine infiltration

INTERVENTIONS:
Drug: tumescent lidocaine infiltration — Tumescent local anesthesia containing dilute lidocaine is infiltrated into subcutaneous tissue prior to liposuction

SUMMARY:
The purpose of this study is to evaluate the effect of lidocaine, delivered into subcutaneous tissue for tumescent local anesthesia, on platelet activation following the tumescent liposuction.

DETAILED DESCRIPTION:
The current research study is intended to examine this hypothesis by determining if tumescent lidocaine increases the results of a test which measures the volume of bleeding which occurs when a tiny standardized incision is made on the forearm. This test is the BA test. The investigators will do BA tests before and after infiltration of lidocaine in the form of tumescent local anesthesia for liposuction and then compare the differences of these BA test results.

The purpose of the present research project is to study how platelet function after surgical trauma (liposuction) is affected by tumescent lidocaine. The investigators hypothesize that lidocaine, delivered in the form of tumescent local anesthesia, inhibits surgical trauma-induced platelet activation as measured by the in-vivo Klein Bleeding Area test (www.onlinePFT).

The Klein Bleeding Area (BA) test is an extension of the classic Ivy Bleeding Time (BT) test. The BT test, an in-vivo test for an abnormal bleeding tendency, involves making a small standardized cut in the skin and measuring the duration of bleeding. The BA test has significantly more sensitivity and specificity than the BT Test.

This research project is a dosage-response clinical trial in which the predictor variable is the milligram per kilogram (mg/kg) dosage of tumescent lidocaine and the response variable is the Bleeding Area (BA). A result indicating that tumescent lidocaine does indeed impair post-operative platelet function would justify a subsequent randomized clinical trial of tumescent lidocaine for preventing post-operative thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have requested tumescent liposuction
* Healthy adults
* ASA Class I, II, or III

Exclusion Criteria:

* Known allergy to lidocaine
* younger than 18 years
* Positive serology for Hepatitis C, HIV
* Chronic fatigue Syndrome
* known bleeding disorder
* significant psychiatric problems
* History of seizures
* Clinically significant cardiac arrhythmia
* Conditions predisposing to surgical site infections
* Active bacterial infection
* taking drugs know to affect hemostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Tumescent lidocaine effects on platelet function following liposuction surgical trauma: a prospective controlled dosage-response phase I clinical trial | two years
  The purpose of the present research project is to study how platelet function after surgical trauma (liposuction) is affected by tumescent lidocaine. We hypothesize that lidocaine, delivered in the form of tumescent local anesthesia, inhibits surgical trauma-induced platelet activation as measured by the in-vivo Klein Bleeding Area test (www.onlinePFT).

CONTACTS AND LOCATIONS:
Locations (1):
- Capistrano Surgicenter, San Juan Capistrano, California, United States